CLINICAL TRIAL: NCT02213211
Title: Impact of a School-based Programme of Malaria Diagnosis and Treatment on School Attendance in Southern Malawi
Brief Title: School-based Programme of Malaria Diagnosis and Treatment in Southern Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Save the Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QA475; 1057 (Other: National Health Sciences Research Committee (NHSRC) Malawi); 6432 (Other: LSHTM ethics reference number)
Record Dates: First submitted 2014-04-07; First posted 2014-08-11 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2014-08

CONDITIONS: Malaria
Keywords: Malawi; Case management; Rapid diagnostic tests; Artemether lumefantrine; School children; School health services; Attendance; Anaemia; Parasitic diseases
MeSH Terms: conditions — Malaria; Anemia; Parasitic Diseases | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diagnosis and treatment of malaria (Experimental): School-based diagnosis and treatment of uncomplicated malaria using malaria RDTs and Artemether lumefantrine as part of Learner Treatment Kits (LTK) used by teachers.
  Drug: Artemether lumefantrine (artemisinin-based combination therapy [ACT], Coartem). Three-day doses of 20mg/120mg, 40mg/240mg, 60mg/360mg and 80mg/480mg Coartem are provided, according to weight, upon a positive rapid diagnostic test (RDT) result.
  Interventions: Drug: Artemether lumefantrine
- No intervention (No Intervention): No intervention provided

INTERVENTIONS:
Drug: Artemether lumefantrine
  Other Names: artemisinin-based combination therapy (ACT); Coartem
  Arms: Diagnosis and treatment of malaria

SUMMARY:
Malaria is an important contributor to ill-health experienced by school-children and may have profound consequences for their learning and educational achievement, and there is a small, but growing, body of evidence that suggests malaria control can help improve educational outcomes. In Malawi, school-aged children are estimated to experience 0.59 clinical attacks of malaria each year, equivalent to 2.1 million attacks among Malawian school-aged children. To avert this health burden and potential education consequences, Save the Children in partnership with the Malawian Ministry of Health is providing treatment of symptomatic malaria cases in schools in southern Malawi, as part of the provision of first aid kits (known as Learner Treatment Kits, LTKs) in schools. To evaluate the impact of this intervention, a cluster randomised trial is being conducted among 58 schools in Traditional Area Chikowi in Malawi, over 12 months. Twenty nine schools are randomly selected to receive LTKs, which include malaria rapid diagnostic tests (RDTs) and artemisinin-based combination therapies (ACTs) to treat uncomplicated malaria, and 29 schools serve as the control group. The primary outcome is school attendance, with secondary outcomes of grade repetition, school drop-out and enrolment as well as morbidity, Plasmodium falciparum infection and anaemia. The study aims to conduct several quantitative and qualitative assessments to help evaluate the external validity of the findings.

DETAILED DESCRIPTION:
This study is a cluster-randomised trial with a comparison group to assess the impact of school-based malaria case management, with malaria rapid diagnostic tests (RDTs) for diagnosis and artemisinin-based combination therapy (ACT) for treatment of uncomplicated malaria incorporated into first aid kits (Learner Treatment Kits) also containing treatment and management for other common minor health issues. A seven day teacher training in the diagnosis and treatment of malaria, other contents of the kit and referral process is provided for the two teachers selected to act as the LTK dispensers in the school, as well as the head teacher. The target population in this study includes children attending the 58 participating primary schools in Traditional Authority Chikowi, Zomba District, Malawi. Twenty nine schools are randomly selected to receive Learner Treatment Kits (LTKs) including RDTs and ACTs to treat uncomplicated malaria, and 29 schools serve as the control group. All children attending schools in the intervention arm have access to the LTK and are eligible for treatment on an opt-out basis, but the accessible study population includes the children randomly selected from classes 2, 4 and 6. The study hypothesis is that that school-based malaria case-management as part of LTKs will reduce rates of absenteeism in Malawian schoolchildren, when compared to those in control schools. The primary outcome is school attendance, with secondary outcomes of grade repetition, school drop-out and enrolment as well as morbidity, Plasmodium falciparum infection and anaemia. The study is designed to provide 80% power to detect a 16% reduction (53% relative reduction) in absenteeism in the intervention group compared to the control group at 5% level of significance. The unit of analysis is the school, but individual-level analysis using suitable generalised linear models, adjusted for clustering by school, will also be undertaken to explore differences in impact of the interventions according to child age, sex, home environment, school quality as well as differences in the uptake of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Student enrolled at participating schools in standards 2, 4 and 6
* Provision of informed consent from parent or guardian
* Provision of assent by student

Exclusion Criteria:

* Student unwilling to participate in the study
* Student known to have a chronic medical condition, which will affect their school attendance

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3667 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
School attendance | 1 year
  School attendance as assessed by class registers and independent spot-checks

SECONDARY OUTCOMES:
Plasmodium falciparum parasitaemia | 1 year
  Presence of malaria parasites in blood sample using microscopy
Anaemia | 1 year
  Anaemia based on haemoglobin concentration assessed using Hemocue photometer
Child wellbeing | 1 year
  Child-recorded wellbeing charts completed by each child three days per week between May and July 2015
Cost effectiveness | 1 year
  Cost effectiveness analysis will consider reductions in absenteeism
Stakeholder perceptions of LTK intervention | End of intervention period
  Perceptions of intervention from teachers, school children and healthcare workers as well as key policy makers obtained through focus group discussions and in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Don P Mathanga, MBBS, Principal Investigator — Malaria Alert Centre, College of Medicine, Malawi; Katherine E Halliday, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Simon J Brooker, DPhil, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Malaria Alert Centre, College of Medicine, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
In order to maximise the usefulness of the study results, it is intended that individual participant data (IPD) will be shared with the wider research community for scientific purposes only, as anonymized, non-personal, individual and summary information. The information will be shared in ways that do not reveal individual participant's identities or household location. The data will be available, on request, through The "Data Compass": the London School of Hygiene & Tropical Medicine (LSHTM) curated digital repository of research data. This will be made available at the stage of publication of the impact results in 2017.

REFERENCES:
- [Result] Mathanga DP, Halliday KE, Jawati M, Verney A, Bauleni A, Sande J, Ali D, Jones R, Witek-McManus S, Roschnik N, Brooker SJ. The High Burden of Malaria in Primary School Children in Southern Malawi. Am J Trop Med Hyg. 2015 Oct;93(4):779-789. doi: 10.4269/ajtmh.14-0618. Epub 2015 Aug 17. PMID 26283750
- [Result] Witek-McManus S, Mathanga DP, Verney A, Mtali A, Ali D, Sande J, Mwenda R, Ndau S, Mazinga C, Phondiwa E, Chimuna T, Melody D, Roschnik N, Brooker SJ, Halliday KE. Design, implementation and evaluation of a training programme for school teachers in the use of malaria rapid diagnostic tests as part of a basic first aid kit in southern Malawi. BMC Public Health. 2015 Sep 17;15:904. doi: 10.1186/s12889-015-2228-x. PMID 26377070
- [Derived] Halliday KE, Witek-McManus SS, Opondo C, Mtali A, Allen E, Bauleni A, Ndau S, Phondiwa E, Ali D, Kachigunda V, Sande JH, Jawati M, Verney A, Chimuna T, Melody D, Moestue H, Roschnik N, Brooker SJ, Mathanga DP. Impact of school-based malaria case management on school attendance, health and education outcomes: a cluster randomised trial in southern Malawi. BMJ Glob Health. 2020 Jan 14;5(1):e001666. doi: 10.1136/bmjgh-2019-001666. eCollection 2020. PMID 32133163
- See also: Social Innovation in Health Initiative (SIHI). This short film forms part of the SIHI case series, showcasing selected social innovations improving healthcare delivery from Africa, Asia and Latin America — http://www.youtube.com/watch?v=MBVzoIk7cFY